CLINICAL TRIAL: NCT02205957
Title: Training Quality in Anesthesia and Intensive Care : Tunisians Residents' Feed Back
Brief Title: Training Quality in Anaesthesia and Intensive Care: Tunisian Residents Feed Back
Status: Completed | Type: Observational
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, Chief of anesthesia department at Mahdia University Hospital, University Hospital, Mahdia
Other Study IDs: Mah2014S1
Record Dates: First submitted 2014-07-26; First posted 2014-08-01 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Training Objectives Achievement
Keywords: anesthesiology and intensive care, quality, training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Training quality: Tunisian residents in anesthesiology and intensive care

SUMMARY:
Opinion survey to assess the level of satisfaction and the expectations of the residents in anesthesiology and intensive care in Tunisia ( North Africa)

DETAILED DESCRIPTION:
The first national anonymous survey to assess the theoretical and practical training quality in anesthesia and intensive care and the improvements propositions.

ELIGIBILITY:
Inclusion Criteria:

* Tunisian nationality
* Resident in anesthesiology and intensive care
* training period : 6 months to four year

Exclusion Criteria:

* training done outside tunisia

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Residents in anesthesiology and intensive care
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
the approval of theoretical and practical teaching | up to four year of training
  A standardized questionnaire assessing the theoretical and practical training was distributed to the 1th,2th,3th and 4th-year anesthesiology residents

SECONDARY OUTCOMES:
Improvement propositions | up to 4th year
  residents can chose from different propositions and give other propositions if not listed in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kolsi Abdessalem, MD, Study Director — Mahdia UNiversity Hospital
Locations (1):
- Mahdia University Hospital, Mahdia, Mahdia Governorate, Tunisia